CLINICAL TRIAL: NCT06979583
Title: Impact of Ureteral Stent Size on the Management of Post Ureteroscopy Pain: a Randomized Single Blind Trial
Brief Title: Impact of Ureteral Stent and Sheaths Size on Post-Operative Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Meghan A. Cooper, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-009000
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Ureteral Stent-Related Symptom; Retrograde Intra-renal Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A: 4.8 Fr Ureteral stents (Experimental)
  Interventions: Device: 4.8 Fr Ureteral stents
- Group B: 7 Fr Ureteral stents (Experimental)
  Interventions: Device: 7 Fr Ureteral stents

INTERVENTIONS:
Device: 4.8 Fr Ureteral stents — After surgery, patients will have the Boston Scientific 4.8 Fr ureteral stent placed.
  Arms: Group A: 4.8 Fr Ureteral stents
Device: 7 Fr Ureteral stents — After surgery, patients will have the Bard 7 Fr ureteral stent placed.
  Arms: Group B: 7 Fr Ureteral stents

SUMMARY:
The purpose of this study is to determine if post-operative stent size impacts stent-related pain and discomfort.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing a retrograde intra-renal surgery (RIRS) (only patients undergoing the procedure for stone treatment will be included) who will require post-operative indwelling ureteral stent placement on a string at the conclusion of the procedure.

Exclusion Criteria:

* Patients with intra-operative ureteral injury who will require ureteral stent for extended time (more than 10 days, in that case a stent without a string will be used).
* Patient undergoing ureteroscopy for any indication other than stone extraction.
* Patients who are currently pregnant as determined by clinical presurgical screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain score post ureteroscopy procedure until stent removal determined by the primary operating team. Stent will be on a string | Starting post-operatively, daily, until stent is removed (estimated 7-14 days)
  Post-operatively, patient will be contacted by study coordinators every day until stent is removed (usually 7-14 days after the surgery) to scale their stent pain on a scale from 1-5 as following: No pain: 1; Mild pain with no need for additional medication: 2; Mild pain with need for additional medication (anticholinergics): 3; Moderate stent pain (requiring narcotics): 4; Severe stent pain (requiring ER visit): 5.

SECONDARY OUTCOMES:
Volume of post-operative correspondence between patients and medical system. | 14 days
  Total number of communications received from patient post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan A. Cooper, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No